CLINICAL TRIAL: NCT03535545
Title: Preliminary Evaluation of [68Ga]CBP8 in Healthy Individuals, Lung Cancer Patients Undergoing Radiation Therapy Prior to the Resection of Locally Advanced Tumors, and Idiopathic Pulmonary Fibrosis Patients
Brief Title: Preliminary Evaluation of [68Ga]CBP8 in Healthy Individuals, Lung Cancer, and Idiopathic Pulmonary Fibrosis Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter Caravan, Professor of Radiology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P002718; R01HL153606 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Fibrosis; Lung Cancer
Keywords: PET Imaging; Molecular Imaging
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Healthy control subjects will be enrolled first and then subjects with lung cancer and idiopathic pulmonary fibrosis and other types of interstitial lung disease or other types of lung disease with a fibrotic component meeting inclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healthy Individuals (Experimental): Healthy volunteers will receive [68Ga]CBP8 and undergo PET imaging.
  Interventions: Drug: [68Ga]CBP8; Diagnostic Test: PET Imaging
- Lung Cancer Subjects (Experimental): Lung cancer patients will receive [68Ga]CBP8 and undergo PET imaging.
  Interventions: Drug: [68Ga]CBP8; Diagnostic Test: PET Imaging
- Pulmonary Fibrosis Subjects (Experimental): Idiopathic pulmonary fibrosis patients or patients with other types of interstitial lung disease with a fibrotic component will receive [68Ga]CBP8 and undergo PET imaging.
  Interventions: Drug: [68Ga]CBP8; Diagnostic Test: PET Imaging
- Subjects with chronic lung allograft dysfunction (CLAD) (Experimental): Subjects with chronic lung allograft dysfunction (CLAD) will receive [68Ga]CBP8 and undergo PET imaging.
  Interventions: Drug: [68Ga]CBP8; Diagnostic Test: PET Imaging
- Subjects with immune-checkpoint-inhibitor (ICI) pneumonitis (Experimental): Subjects with immune-checkpoint-inhibitor (ICI) pneumonitis will receive [68Ga]CBP8 and undergo PET imaging.
  Interventions: Drug: [68Ga]CBP8; Diagnostic Test: PET Imaging

INTERVENTIONS:
Drug: [68Ga]CBP8 — Up to 15 mCi of [68Ga]CBP8 will be administered to each subject.
Diagnostic Test: PET Imaging — All subjects will undergo PET imaging after administration of [68Ga]CBP8.

SUMMARY:
The goal of this study is to investigate the safety of [68Ga]CBP8 and its efficacy to detect collagen deposition in pulmonary fibrosis.

DETAILED DESCRIPTION:
The investigators have developed [68Ga]CBP8, a gallium-68 labeled collagen binding PET imaging probe, which selectively binds collagen type I. Collagen deposition is a pivotal event in several human conditions including pulmonary fibrosis. The investigator's studies in mice showed that [68Ga]CBP8 binds collagen with high affinity and has excellent pharmacological and pharmacokinetic profiles with high target uptake and low retention in background tissues and organs. [68Ga]CBP8 was shown in a mouse model to be effective for detecting lung fibrosis. [68Ga]CBP8 showed high specificity for pulmonary fibrosis and high target:background ratios in diseased animals. In addition, [68Ga]CBP8 could be used to monitor response to treatment. Ex vivo analysis of lung tissue from patients with IPF supported the animal findings.

The investigators thus aim to perform the first in human studies of [68Ga]CBP8:

1. To evaluate the safety of [68Ga]CBP8 and its whole body distribution, metabolism, pharmacokinetics, and radiation burden in healthy volunteers.
2. To establish the accuracy of [68Ga]CBP8-PET to detect radiation-induced fibrosis in lung cancer patients and correlate collagen-targeted [68Ga]CBP8-PET imaging with HRCT and histology in lung cancer patients.
3. To determine whether collagen deposition as assessed by [68Ga]CBP8-PET molecular imaging can predict disease progression in IPF patients and patients with other types of ILD with a fibrotic component.

ELIGIBILITY:
Inclusion Criteria: Total enrollment for all groups will not exceed 100 subjects.

* Group 1: Healthy subjects
* Age greater than 18 years
* Be deemed healthy at screening visit as determined by the physician investigator or nurse practitioner, based on the following assessments at Screening: physical examination, medical history, and vital signs
* Have the ability to give written informed consent;
* No known history of pulmonary disease (excluding pulmonary nodules);
* No prior history of tobacco use.

Group 2: Lung cancer subjects

* Eligible patients will be those harboring locally advanced clinical stage IIIA NSCLC who are deemed candidates for multi-modality therapy, i.e. concurrent chemotherapy and radiation followed by pulmonary resection.
* Age greater than 18 years
* Have the ability to give written informed consent.
* No tobacco use within the prior 6 months.

Group 3: Subjects with pulmonary fibrosis

* IPF (with a UIP or probable UIP pattern); or other forms of interstitial lung disease (ILD), including CTD-ILD, with a fibrotic component as noted by the presence of reticular markings and / or traction bronchiectasis and / or honeycombing on CT;
* Age: 40-80 years old;
* Have the ability to give written informed consent;
* No tobacco use within the prior 6 months

Group 4: Subjects with chronic lung allograft dysfunction (CLAD)

* Status post lung transplantation
* Clinical diagnosis of chronic lung allograft dysfunction
* Age: 40-80 years old;
* Have the ability to give written informed consent;
* No tobacco use within the prior 6 months

Group 5: Subjects with immune-checkpoint-inhibitor (ICI) pneumonitis

* CT findings with ground glass opacities / consolidation or fibrotic changes with new onset during or within 3 months of receipt of ICI therapy
* Age greater than 18 years
* Have the ability to give written informed consent
* No tobacco use within the prior 6 months

Exclusion Criteria:

* Electrical implants such as cardiac pacemaker or perfusion pump;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing;
* eGFR of less than 30 mL/min/1.73 m2 within the past 90 days for group 4 subjects; history of chronic kidney disease for subjects in groups 1-3 and 5;
* Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test is required for females having child-bearing potential before the subject can participate);
* Claustrophobic reactions;
* Research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Unable to lie comfortably on a bed inside the MR-PET;
* BMI > 33 (limit of the MRI table);
* Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures);
* Known history of pulmonary disease (except for pulmonary fibrosis in the study group, ICI pneumonitis in the study group, or CLAD in the study group), recent pneumonia or respiratory tract infections within 6 weeks of enrollment, prior radiation therapy to the thorax (except for the lung cancer patients in aim 2);
* Pneumonia or other acute respiratory illness within 6 weeks of study entry (except for pulmonary fibrosis), pneumonia defined with elevated WBC, fever, infiltrate on CXR and need for antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability to detect increased collagen deposition in pulmonary fibrosis. | Two hours
  Probe lung uptake will be measured in pulmonary fibrosis subjects and compared to lung uptake in healthy volunteers. We expect greater uptake in the lungs of IPF patients and patients with other types of ILD with a fibrotic component.

SECONDARY OUTCOMES:
Ability of the degree of collagen deposition to predict disease progression. | Up to 36 months
  Probe lung uptake in pulmonary fibrosis patients will be correlated with change in forced vital capacity over the prior 12 months and prospectively over the following 12-36 months.

OTHER OUTCOMES:
Ability of [68Ga]CBP8 to detect collagen deposition in areas of radiation injury. | Up to 3 months
  Probe lung uptake will be measured in lung cancer patients prior to surgical resection and compared to histologic measures of fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B Montesi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537
- [Background] Desogere P, Tapias LF, Rietz TA, Rotile N, Blasi F, Day H, Elliott J, Fuchs BC, Lanuti M, Caravan P. Optimization of a Collagen-Targeted PET Probe for Molecular Imaging of Pulmonary Fibrosis. J Nucl Med. 2017 Dec;58(12):1991-1996. doi: 10.2967/jnumed.117.193532. Epub 2017 Jun 13. PMID 28611243
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Izquierdo-Garcia D, Desogere P, Fur ML, Shuvaev S, Zhou IY, Ramsay I, Lanuti M, Catalano OA, Catana C, Caravan P, Montesi SB. Biodistribution, Dosimetry, and Pharmacokinetics of 68Ga-CBP8: A Type I Collagen-Targeted PET Probe. J Nucl Med. 2023 May;64(5):775-781. doi: 10.2967/jnumed.122.264530. Epub 2022 Dec 8. PMID 37116909
- [Derived] Abston E, Zhou IY, Saenger JA, Shuvaev S, Akam E, Esfahani SA, Hariri LP, Rotile NJ, Crowley E, Montesi SB, Humblet V, Arabasz G, Catana C, Fintelmann FJ, Caravan P, Lanuti M. Noninvasive Quantification of Radiation-Induced Lung Injury using a Targeted Molecular Imaging Probe. medRxiv [Preprint]. 2023 Sep 26:2023.09.25.23295897. doi: 10.1101/2023.09.25.23295897. PMID 37808864